CLINICAL TRIAL: NCT00965705
Title: Dialectical Behavior Therapy for Early Non-Responders to CBT
Brief Title: Stepped Care Treatment for Binge-Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eunice Chen, Study Principal Investigator, Temple University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20472; K23MH081030-01 (NIH)
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Binge Eating Disorder
Keywords: Binge Eating Disorder; overeating; binge eating; women; overweight; compulsive overeating
MeSH Terms: conditions — Binge-Eating Disorder; Hyperphagia; Bulimia; Overweight | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Guided Self Help (Active Comparator)
  Interventions: Behavioral: Therapy
- Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Therapy
- Dialectical Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Therapy

INTERVENTIONS:
Behavioral: Therapy — Individual Therapy and Group Therapy

SUMMARY:
Temple University is looking for women to participate in a study to evaluate the treatment options available to women living with binge eating disorder.

Binge-Eating Disorder is a significant public health problem for women. Despite this, there is limited research on how best to treat this disorder at varying levels of severity. The purpose of this NIMH-funded study is to enroll individuals in a brief form of cognitive-behavior therapy. If more intense treatment is needed, individuals will be randomly assigned to more intensive group and individual treatments (Cognitive-Behavior Therapy or Dialectical Behavior Therapy). Both of these treatments are talking therapies that have been adapted for women living with binge-eating disorder and are free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Adult female, 18 years to 60 years
* Meets DSM-IV criteria for Binge Eating Disorder
* Resides within commuting distance
* Consents to research protocol, i.e.
* 18-24 months in assessment and treatment
* willing to be part of a biological assessment/physiological assessment
* have to be prepared that they will receive a brief individual treatment and if this does not work for them, that they will receive more intensive treatment including both group and individual treatment.
* agreement not to see other health professionals unless recommended
* seeing their own Primary care Physician/Nurse Practitioner for medical screening prior to study (i.e., before being allocated a guided self-help therapist)
* payment for their own medical assessment, monitoring, and medication if needed

Exclusion Criteria:

* Anorexia nervosa
* Schizophrenia, Schizophreniform, or Schizoaffective Disorders, Psychosis NOS, or Bipolar Mood Disorder
* Needs priority treatment for other debilitating conditions, e.g. current substance dependence requiring inpatient detox
* chronic absence of shelter
* IQ less than 70
* Impending jail/prison, court order to treatment, court order to treatment or to jail, or agency order to treatment or to loss of child custody (due to consequent inability to freely drop-out of treatment)
* Is pregnant, plans to become pregnant during treatment, or becomes pregnant before random assignment to study condition
* Medical instability
* Has had or is seeking Gastric bypass surgery
* On anti-seizure medication, beta-blockers, asthma medication, medication for heart disease, or any other medication that affects appetite or weight
* Psychotropics are acceptable if the doses are stable for at least 3 months prior to screening

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of objective binge eating days or objective binge eating frequency using the Eating Disorders Examination-16 over the last month | Up to 12 months after randomization
  Number of objective binge eating days or objective binge eating frequency using the Eating Disorders Examination-16 over the last month

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Y Chen, PHD, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Chen EY, Cacioppo J, Fettich K, Gallop R, McCloskey MS, Olino T, Zeffiro TA. An adaptive randomized trial of dialectical behavior therapy and cognitive behavior therapy for binge-eating. Psychol Med. 2017 Mar;47(4):703-717. doi: 10.1017/S0033291716002543. Epub 2016 Nov 17. PMID 27852348
- [Result] Southward MW, Christensen KA, Fettich KC, Weissman J, Berona J, Chen EY. Loneliness mediates the relationship between emotion dysregulation and bulimia nervosa/binge eating disorder psychopathology in a clinical sample. Eat Weight Disord. 2014 Dec;19(4):509-13. doi: 10.1007/s40519-013-0083-2. PMID 24235091
- See also: Temple University Eating Disorders (TED) Website — http://sites.temple.edu/tedp